CLINICAL TRIAL: NCT01429441
Title: A Randomized, Sham-controlled, Double-masked, Multicenter Study Evaluating Ocriplasmin Treatment for Symptomatic Vitreomacular Adhesion Including Macular Hole
Brief Title: Ocriplasmin for Treatment for Symptomatic Vitreomacular Adhesion Including Macular Hole
Acronym: OASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-MV-014
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-01

CONDITIONS: Vitreomacular Adhesion Including Macular Hole
MeSH Terms: interventions — microplasmin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ocriplasmin (Experimental)
  Interventions: Drug: Ocriplasmin
- Sham injection (Sham Comparator)
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Ocriplasmin — 0.125 mg single intravitreal injection
  Arms: Ocriplasmin
Other: Sham injection — Sham injection
  Arms: Sham injection

SUMMARY:
The purpose of this study is to evaluate the treatment of symptomatic vitreomacular adhesion / (VMT) including macular hole with ocriplasmin.

DETAILED DESCRIPTION:
The present study is designed to assess anatomical and functional outcomes following a single intravitreal injection of ocriplasmin 0.125mg in subjects with symptomatic vitreomacular adhesion (VMA)/ (VMT) including macular hole.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older and of either gender
* Presence of vitreomacular adhesion
* Best corrected visual acuity (BCVA) of 20/32 or worse in study eye
* BCVA of 20/800 or better in the non-study eye

Exclusion Criteria:

* History or current evidence of proliferative retinopathy, exudative age-related macular degeneration (AMD) or retinal vein occlusion in the study eye
* Any vitreous hemorrhage or any other vitreous opacification which precludes the visualization of the posterior pole by visual inspection OR adequate assessment of the macula by spectral-domain optical coherence tomography (SD-OCT) in the study eye
* Macular hole of > 400 µm diameter in the study eye
* Presence of epiretinal membrane (ERM)
* Aphakia in the study eye
* High myopia (more than 8D) in study eye
* History of rhegmatogenous retinal detachment in either eye
* History of vitrectomy in the study eye
* Previous participation in this trial or prior administration of ocriplasmin in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Consultants Medical Group, Sacramento, California
  - West Coast Retina Group, Inc, San Francisco, California
  - Bay Area Retina Associates, Walnut Creek, California
  - MedEye Associates, Miami, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Sabates Eye Center Research, Kansas City, Missouri
  - Eyesite Opthalmic Services, PA, Portsmouth, New Hampshire
  - Retina-Vitreous Center, PA, New Brunswick, New Jersey
  - Retina Association of NJ, Teaneck, New Jersey
  - Retina Vitrous Surgeons of CNY, Syracuse, New York
  - Southeast Clinical Research, PA, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Mid Atlantic Retina, Huntingdon Valley, Pennsylvania
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants, PA, Fort Worth, Texas
  - Vitroretinal Consultants, Houston, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Retina Consultants of San Antonio, San Antonio, Texas
  - Eye Care Associate, Tyler, Texas

REFERENCES:
- [Derived] Velaga SB, Nittala MG, Ip MS, Duchateau L, Sadda SR. Post hoc analysis of ellipsoid zone changes beyond the central subfield in symptomatic vitreomacular adhesion patients from the OASIS trial. BMJ Open Ophthalmol. 2021 Jun 21;6(1):e000648. doi: 10.1136/bmjophth-2020-000648. eCollection 2021. PMID 34250257
- [Derived] Yu TM, Dugel PU, Haller JA, Kaiser PK, Arnold RJ. Budget impact analysis of ocriplasmin for the treatment of symptomatic vitreomacular adhesion in the USA. J Comp Eff Res. 2018 Dec;7(12):1195-1207. doi: 10.2217/cer-2018-0057. Epub 2018 Oct 23. PMID 30350717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 25 study sites in the United States. The first subject was enrolled on 02 November 2011 and the last subject completed the study on 22 October 2014.
Groups:
- Ocriplasmin: Subjects in the ocriplasmin group received a single intravitreal injection of ocriplasmin 0.125mg
- Sham: Subjects in the sham group received a single sham injection
Period: Overall Study
Arm/Group | Ocriplasmin | Sham
Started | 146 | 74
Completed | 108 | 51
Not Completed | 38 | 23
Not completed — Adverse Event | 5 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 27 | 18

BASELINE CHARACTERISTICS:
Population: Safety Set: The Safety Set consists of all subjects who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin | Sham | Total
Number analyzed (Participants) | 146 | 74 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.99) | 68.5 (10.94) | 69.1 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 45 | 148
  Male | 43 | 29 | 72

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Pharmacological Vitreomacular Adhesion (VMA) / (Vitreomacular Traction [VMT]) Resolution at Day 28
Description: Pharmacological VMA resolution without anatomical defect, based on SD-OCT and determined by the masked central reading center (CRC), with post-resolution vitrectomy considered as a failure. Missing data were imputed using the last observation carried forward (LOCF) method.
Time Frame: Day 28
Population: Full Analysis Set (FAS): The FAS is the set of all randomized subjects who received the initial treatment, and for whom data of at least 1 post-injection efficacy assessment was present. Two (2) subjects (1 in each treatment group) were excluded from the FAS as they withdrew consent and did not attend any of the post-injection visits.
Measure: Number (95% Confidence Interval); unit: Percentage (weighted across strata)
Arm/Group | Ocriplasmin | Sham
Number analyzed (Participants) | 145 | 73
Percentage (weighted across strata) | 41.7 [33.7 to 49.8] | 6.2 [0.9 to 11.6]

2. Secondary Outcome: Proportion of Subjects With a ≥2 Lines Improvement in Best-corrected Visual Acuity (BCVA) From Baseline at Month 24
Description: ≥2 lines improvement in BCVA from baseline, irrespective of vitrectomy. Missing data were imputed using the LOCF method.
Time Frame: Month 24
Population: FAS. 1 subject did not have BCVA results at baseline and was excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage (weighted across strata)
Arm/Group | Ocriplasmin | Sham
Number analyzed (Participants) | 144 | 73
Percentage (weighted across strata) | 50.5 [42.4 to 58.5] | 39.1 [28.3 to 49.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the injection day (Day 0) up to discontinuation from the study or completion of the study (Month 24).
Description: The Safety Set consisted of all subjects who received study treatment and was used for all safety analyses. All subjects were included in the Safety Set: 146 subjects in the ocriplasmin group and 74 subjects in the sham group.
Arm/Group | Ocriplasmin | Sham
Serious Adverse Events (participants affected / at risk) | 49/146 | 27/74
Other Adverse Events (participants affected / at risk) | 132/146 | 57/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=146) | Sham (N=74)
Macular hole (Eye disorders) | 21 (21) | 9 (9)
Retinal detachment (Eye disorders) | 3 (3) | 1 (1)
Vitreous adhesions (Eye disorders) | 2 (2) | 2 (2)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Night blindness (Eye disorders) | 1 (1) | 0 (0)
Pupillary reflex impaired (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 2 (2)
Retinal toxicity (Eye disorders) | 1 (1) | 0 (0)
Retinal vasculitis (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3)
Intraocular pressure increased (Investigations) | 3 (3) | 2 (4)
Retinogram abnormal (Investigations) | 1 (1) | 0 (0)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myelomonocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adrenalectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=146) | Sham (N=74)
Vitreous floaters (Eye disorders) | 57 (75) | 6 (6)
Photopsia (Eye disorders) | 44 (53) | 6 (7)
Vision blurred (Eye disorders) | 28 (34) | 4 (6)
Cataract nuclear (Eye disorders) | 23 (30) | 10 (11)
Cataract (Eye disorders) | 22 (26) | 10 (10)
Macular fibrosis (Eye disorders) | 22 (26) | 8 (8)
Visual acuity reduced (Eye disorders) | 22 (25) | 18 (26)
Visual impairment (Eye disorders) | 21 (38) | 4 (6)
Eye pain (Eye disorders) | 20 (22) | 6 (10)
Photophobia (Eye disorders) | 19 (22) | 0 (0)
Posterior capsule opacification (Eye disorders) | 17 (20) | 3 (4)
Subretinal fluid (Eye disorders) | 17 (18) | 4 (4)
Chromatopsia (Eye disorders) | 16 (18) | 2 (3)
Conjunctival hemorrhage (Eye disorders) | 15 (17) | 2 (2)
Metamorphopsia (Eye disorders) | 14 (15) | 5 (6)
Retinal hemorrhage (Eye disorders) | 12 (12) | 4 (7)
Retinal pigment epitheliopathy (Eye disorders) | 11 (12) | 3 (3)
Macular hole (Eye disorders) | 9 (9) | 1 (1)
Ocular discomfort (Eye disorders) | 9 (10) | 2 (2)
Cystoid macular edema (Eye disorders) | 8 (10) | 2 (2)
Lacrimation increased (Eye disorders) | 8 (10) | 2 (3)
Foreign body sensation in eyes (Eye disorders) | 5 (5) | 6 (6)
Retinal tear (Eye disorders) | 2 (2) | 4 (5)
Cataract cortical (Eye disorders) | 1 (1) | 4 (4)
Color vision tests abnormal (Investigations) | 43 (89) | 14 (18)
Ophthalmological examination abnormal (Investigations) | 29 (44) | 15 (21)
Intraocular pressure increased (Investigations) | 10 (10) | 9 (11)
Visual acuity tests abnormal (Investigations) | 9 (10) | 2 (2)
Hypertension (Vascular disorders) | 10 (12) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 4 (4)
Sinusitis (Infections and infestations) | 8 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have the right to the 1st publication of the Study results (joint, multi-center publication in conjunction with PI). Following the 1st publication, PI may publish data/results from the Study; provided that PI submits the proposed publication to Sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may request that Confidential/Proprietary Information be deleted and/or publication be postponed to protect Sponsor's intellectual property rights.